CLINICAL TRIAL: NCT00149357
Title: Determining the Risk of Fetal Loss in Women With Unprovoked Venous Thromboembolism (VTE) Who Do NOT Have Identifiable Inherited Thrombophilia Compared With Women Who Have the Diagnosis of VTE Excluded
Brief Title: Fetal Loss in Women With Unprovoked Thromboembolism (FLUTE)
Status: Terminated | Type: Observational
Why Stopped: Funding withdrawn due to low enrollment
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CTMG-2005-FLUTE
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Venous Thromboembolism; Fetal Death
Keywords: venous thromboembolism; VTE; thrombophilia; fetal loss
MeSH Terms: conditions — Venous Thromboembolism; Fetal Death; Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1, 2 ,3: Group 1 Women with unprovoked VTE and No Known Thrombophilia Group 2 Women who are investigated for VTE and are negative (Control) Group 3 Women with unprovoked VTE who have Thrombophilia
  Interventions: Other: Thrombophilia Testing

INTERVENTIONS:
Other: Thrombophilia Testing — TP testing in Group 1 and 3 only

SUMMARY:
The purpose of this study is to determine the risk of fetal loss in women with unprovoked venous thromboembolism (VTE) who do not have identifiable inherited thrombophilia compared with women who have the diagnosis of venous thromboembolism (VTE) excluded.

ELIGIBILITY:
Inclusion Criteria:

* Female
* At least 18 years of age
* Symptomatic for unprovoked venous thromboembolism (deep vein thrombosis [DVT] or pulmonary embolism [PE])
* At least one pregnancy not terminated intentionally

Exclusion Criteria:

* Previous VTE in patients with current VTE excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huyen Tran, M.D., Study Chair — McMaster University; Department of Medicine; Jeffrey Ginsberg, M.D., Principal Investigator — McMaster University; Department of Medicine; Clive Kearon, M.D., Principal Investigator — McMaster University; Department of Medicine; Jim Julian, M.Math, Principal Investigator — McMaster University; Dept. of Clinical Epidemiology & Biostatistics; Val Mueller, M.D., Principal Investigator — McMaster University; Division of Obstetrics and Gynecology
Locations (5):
- Monash Medical Centre, Clayton, Victoria, Australia
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Henderson Research Centre, Hamilton, Ontario